CLINICAL TRIAL: NCT03818282
Title: Efficacy and Safety of Paclitaxel for Injection (Albumin-bound) in Combination With Carboplatin for First-line Chemotherapy of Ovarian Cancer: A Multicenter, Open-label, Single-arm Phase 2 Clinical Study
Brief Title: Efficacy and Safety of Paclitaxel for Injection (Albumin-bound) for First-line Chemotherapy of Ovarian Cancer
Acronym: OC-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ding Ma, Director, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-GYN/OC-01
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel for injection (albumin-bound) (Experimental)
  Interventions: Drug: Paclitaxel for injection (albumin-bound)

INTERVENTIONS:
Drug: Paclitaxel for injection (albumin-bound) — Paclitaxel for injection (albumin-bound) 260 mg/m2, i.v., d1; AUC = 5 for carboplatin injection, i.v., infusion completed on day 1-3; Repeated every 3-4 weeks for 6-8 cycles.

SUMMARY:
Preliminary evaluation of the efficacy and safety of paclitaxel for injection (albumin-bound) in combination with carboplatin for first-line chemotherapy of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years;
* Histologically confirmed epithelial ovarian cancer, fallopian tube cancer and primary peritoneal cancer;
* Patients with stage IC-IV according to the International Federation of Obstetrics and Gynecology (FIGO) and who underwent an ideal tumor reduction procedure within 6 weeks prior to enrollment;
* Lesion is measurable according to RECIST 1.1 criteria or patient's CA125 is evaluable according to GCIG criteria;
* ECOG performance status of 0-2;
* Expected survival ≥ 3 months;
* Bone marrow function: Neutrophils ≥ 1.5×109/L, platelets ≥ 100×109/L, hemoglobin ≥ 90 g/L;
* Hepatic and renal function: Serum creatinine ≤ 1.5×ULN; AST and ALT ≤ 1.5×ULN or ≤ 5×ULN in the presence of hepatic metastasis; Total bilirubin ≤ 1.5×ULN, or ≤ 2.5×ULN in patients with Gilbert's syndrome;
* Must agree to use effective contraception during the trial; Women of childbearing potential must have a negative serum or urine pregnancy test; Non-lactating patients.

Exclusion Criteria:

* Ovarian low-grade malignant tumor patients;
* Patients who have received abdominal or pelvic radiotherapy;
* Patients with central nervous system disease or brain metastases;
* Other malignancies have occurred within the last 5 years, except for cervical carcinoma in situ, non-melanoma skin cancers that have been cured;
* Prior Grade ≥ 2 sensory or motor neuropathy;
* Uncontrolled serious medical conditions that, in the opinion of the investigator, would affect the ability of the subject to receive the study regimen, such as concomitant serious medical conditions, including severe heart disease, cerebrovascular disease, uncontrolled diabetes mellitus, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.;
* Known to be hypersensitive, highly sensitive, or intolerant to study-related medications or their excipients;
* Receive other study drug chemotherapy within 30 days of the first dose of chemotherapy;
* Patients not suitable for participation in this study judged by investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free Survival | 2 year
  PFS